CLINICAL TRIAL: NCT00603031
Title: Effect of GLP-1 and GIP on the Maximal Insulin Secretory Capacity in Type-1 Diabetes Mellitus
Brief Title: Effect of GLP-1 and GIP on Insulin Secretion in Type-1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Urd Kielgast,MD, Urd Kielgast, MD
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H-D-2007-0076; 2008-000305-11 (Other: Ethical Comitee, Copenhagen, Denmark)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2009-08

CONDITIONS: Type-1 Diabetes Mellitus
MeSH Terms: interventions — Glucagon-Like Peptide 1; Incretins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLP-1 (Experimental): time -30-90 min: Continuous infusion with GLP-1 (1,2pmol/kg/min) time 0-90 min:hyperglycemic clamp(20mmol/L) time 45 min:infusion of L-Arginine (5g).
  Interventions: Other: glucagon like peptide -1
- NaCl (Placebo Comparator): time -30-90 min: Continuous infusion with NaCl time 0-90 min:hyperglycemic clamp(20mmol/L) time 45 min:infusion of L-Arginine (5g).
  Interventions: Other: NaCl
- GIP (Experimental): time -30-90 min: Continuous infusion with GIP-1 (3,6pmol/kg/min) time 0-90 min:hyperglycemic clamp(20mmol/L) time 45 min:infusion of L-Arginine (5g).
  Interventions: Other: glucose dependent insulinotropic polypeptide

INTERVENTIONS:
Other: glucagon like peptide -1 — continuous infusion 1,2 pmol pr. kg pr minute at 120 minutes
  Arms: GLP-1
Other: NaCl — infusion with NaCl for 120 minutes as placebo-arm
  Arms: NaCl
Other: glucose dependent insulinotropic polypeptide — continuous infusion with GIP-1 (3,6pmol/kg/min) at 120 minutes.
  Arms: GIP

SUMMARY:
study hypothesis: treatment with GLP-1 and/or GIP is able to potentiate the maximal stimulated insulin secretion even in c-peptide negative type-1 diabetic patients classified as having no residual beta cell function left.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Type-1 diabetes diagnosed between 5-40 years of age
* Normal weight(BMI 18-27),
* Insulin treatment from time of diagnosis.

Exclusion Criteria:

* Severe complications to diabetes
* Abnormal liver or kidney function
* Haemoglobin below the lower limit
* Macroalbuminuria
* Systemic disease
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
phase insulin response and phase insulin response measured as incremental area under the curve from 0-10 minutes and incremental area under the curve from 10-45 minutes respectively after iv glucose | 2 hours

SECONDARY OUTCOMES:
maximal insulin response defined as mean insulin at time 47 and 49 minutes (2 and 4 minutes after infusion of L-Arginine) | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Urd Kielgast, MD, Principal Investigator — unafilliated
Locations (1):
- Dept. of Endocrinology, Hvidovre Hospital, Copenhagen, Denmark